CLINICAL TRIAL: NCT07290257
Title: Long-Term Low-Intervention SafEty and Clinical Outcomes Clinical Study of LivmArli® in Patients With Alagille Syndrome in the European Union (LEAP-EU)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MRX-803
Record Dates: First submitted 2025-09-17; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Alagille Syndrome
Keywords: ALGS; Liver Diseases; Alagille Syndrome; Livmarli; Maralixibat; Cholestasis; Pruritus; Itching; IBAT inhibitor
MeSH Terms: conditions — Alagille Syndrome; Liver Diseases; Cholestasis; Pruritus | interventions — maralixibat

STUDY DESIGN:
Intervention Model Description: The study will enroll a primary cohort with a minimum of 45 previously untreated (treatment naïve) patients with ALGS including at least 5 participants <1 year of age, 30 participants between 1 and 5 years of age, and 10 participants >5 years of age. A supplemental cohort of participants who have previously received Livmarli will also be enrolled. There is no enrollment limit for supplementary cohort. For admin purposes, the number has been set to 55 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Alagile Syndrome treated with Livmarli (Experimental): Primary cohort with a minimum of 45 previously untreated (treatment naïve). Supplemental cohort of participants who have previously received Livmarli.
  Interventions: Drug: Livmarli Oral Product

INTERVENTIONS:
Drug: Livmarli Oral Product — Participants will be treated according to standard of care for the duration of the study and Schedule of Assessments.
  Other Names: Maralixibat

SUMMARY:
The key objectives of this low-intervention clinical study are to evaluate tolerability, long-term safety and long-term efficacy for patients with Alagille syndrome (ALGS) who are prescribed Livmarli.

DETAILED DESCRIPTION:
This is a multicenter, open-label, low-intervention clinical study in participants diagnosed with Alagille syndrome (ALGS) who are treated with Livmarli for cholestatic pruritus.

Participants will be treated according to standard of care for the duration of the study and Schedule of Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and assent (as applicable)
* ≥2 months of age at Day 1
* A clinically and/or genetically confirmed ALGS diagnosis with pruritus secondary to chronic cholestasis
* For the primary cohort, prescribed Livmarli at time of study entry
* For the supplemental cohort, prescribed Livmarli prior to study entry

Exclusion Criteria:

* History of Liver Transplant
* Any contraindications against Livmarli (as per SmPC)
* Any condition or abnormality that, in the opinion of the investigator, may interfere with the participation in or completion of the study
* Received an investigational drug within 30 days before the first dose of Livmarli (Participation in previous maralixibat studies or expanded-access programs is acceptable.)
* Baseline data before start of treatment of Livmarli are unavailable (<2 values before treatment) for key safety (LFTs, FSV laboratory results) and key efficacy (sBA, pruritus) parameter

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2030-09-22 (Estimated); Study Completion 2030-12-22 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to 7 days after the last dose of Livmarli.
  Number and proportion of participants with AEs.
Liver function tests (LFTs) - measuring enzyme activity or concentration | Once every 3-4 months, for 5 years.
  Change in LFTs from Baseline: Total and direct bilirubin, aminotransferases, GGT, and alkaline phosphatase.
Fat-Soluble Vitamins (FSV) Concentration | Once every 3-4 months, for 5 years.
  Change in FSV levels (vitamins A, D, and E) from Baseline.
International Normalized Ratio (INR) | Once every 3-4 months, for 5 years.
  Change in INR level from Baseline.
Long-Term Clinical Outcomes | Once every 3-4 months, for 5 years.
  Number of participants with surgical biliary diversion, liver transplantation, liver transplant waitlist status change, clinically evident portal hypertension, complications of liver cirrhosis, liver carcinoma, liver decompensation, and death.

CONTACTS AND LOCATIONS:
Locations (13):
- Belgium (2):
  - Cliniques Universitaires Saint Luc (UCLouvain), Brussels
  - University Hospital Gent (UZ Gent), Ghent
- France (3):
  - Hospices Civils de Lyon - Hopital Femme Mère Enfant, Bron, Auvergne-Rhône-Alpes
  - CHU de Toulouse - Hôpital des Enfants, Toulouse, Occitanie
  - Bicetre University Hospital, Le Kremlin-Bicêtre, Île-de-France Region
- Germany (3):
  - Charite Berlin, Berlin
  - Children's University Hospital Essen, Essen
  - University Hospital Hamburg-Eppendorf, Hamburg
- Italy (2):
  - AO Ospedale PAPA GIOVANNI XXIII, Bergamo, Lombardy
  - Istituto mediterraneo trapianti - ISMETT, Palermo, Sicily
- University Medical Center Groningen (UMCG), Groningen, Netherlands
- Spain (2):
  - Hospital Universitairo Vall D'Hebron, Barcelona, Catalonia
  - Hospital Universitario La Paz, Madrid